CLINICAL TRIAL: NCT03514706
Title: The Ultrasound Estimation of Extravascular Lung Water in Volume Controlled Versus Pressure Controlled Ventilation After One Lung Ventilation in Thoracoscopic Surgery. A Comparative Study
Brief Title: Effect of PCV and VCV on Extravascular Lung Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hisham Hosny, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: AnesthN-8-2018
Record Dates: First submitted 2018-04-02; First posted 2018-05-02 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Extravascular Lung Water
Keywords: Extravascular lung water; one lung ventilation; volume controlled ventilation; pressure controlled ventilation

STUDY DESIGN:
Intervention Model Description: Adult patients scheduled for elective thoracic surgery with one lung ventilation will be included in the study. Patients will be randomly allocated into one of two groups:
  Group V: will receive volume controlled mechanical ventilation. Group P: will receive pressure controlled mechanical ventilation.
Who Masked: Investigator
Masking Description: Lung ultrasound will be done by an investigator blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volume controlled ventilation (Experimental): Group V: Patients will receive volume controlled mechanical ventilation. (Vt 7ml/kg ideal body weight).
  Interventions: Diagnostic Test: volume controlled ventilation
- Pressure controlled ventilation (Experimental): Group P: Patients will receive pressure controlled mechanical ventilation. (to achieve Vt 7 ml/kg ideal body weight, Pmax 30 cmH2O)
  Interventions: Diagnostic Test: pressure controlled ventilation

INTERVENTIONS:
Diagnostic Test: volume controlled ventilation — Lung ultrasound (LUS) will be performed with a 2-4 MHz phased array probe. Patients will be scanned in supine position by a recording 5 seconds videos. LUS will be assessed for the presence of B lines.
  The sum of lung comets produces a score reflecting the extent of lung water accumulation. LUS will be obtained by scanning 12-rib interspaces. The sum of B-lines on each scanning site yields a score from 0 to 36
  Other Names: LUS
  Arms: Volume controlled ventilation
Diagnostic Test: pressure controlled ventilation — Lung ultrasound (LUS) will be performed with a 2-4 MHz phased array probe. Patients will be scanned in supine position by a recording 5 seconds videos. LUS will be assessed for the presence of B lines.
  The sum of lung comets produces a score reflecting the extent of lung water accumulation. LUS will be obtained by scanning 12-rib interspaces. The sum of B-lines on each scanning site yields a score from 0 to 36
  Other Names: LUS
  Arms: Pressure controlled ventilation

SUMMARY:
Volume controlled ventilation (VCV) and pressure controlled ventilation (PCV) are the common ventilatory modes during OLV undergoing thoracic surgery. A controversy regarding which ventilation mode is better for oxygenation during OLV with PCV enhances oxygenation more than VCV ;given its initial high peak inspiratory flow rates and its rapidly decelerating flow pattern. However, this high peak inspiratory flow rate might also provoke lung injury via shearing and traction forces on the alveoli. Extravascular lung water describes water within the lungs but outside pulmonary vasculature. Lung ultrasound (LUS) assessment of EVLW by B-lines provides a reliable and easy alternative.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged (18-60 years), undergoing elective thoracoscopic surgery with one lung ventilation

Exclusion Criteria:

* Emergency surgeries.
* Left Ventricular ejection fraction less than 40%.
* Any patient known to have pulmonary hypertension
* Patients with preoperative congestive heart failure, cardiogenic shock, preoperative pulmonary edema
* Hepatic patients (liver functions double the upper reference range)
* Morbid obesity (BMI > 40).
* Renally impaired patients with creatinine more than 2 mg/dl.
* Any patient with respiratory dysfunction (FEV1<60% of the expected).
* Any patient with previous thoracic surgery.
* One lung ventilation more than 2 hours

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Lung ultrasound score | change of lung ultrasound scores introperatively during double lung and single lung ventilation and after 2 hours postoperatively compared to baseline scores before anesthesia induction
  The sum of B lines reflects the extent of lung water accumulation. The lung ultrasound score(LUS) will be obtained by scanning 12-rib interspaces. The dependent lung will be divided into six areas: two anterior areas, two lateral areas, and two posterior areas. The anterior chest wall (zone 1) will be delineated from the parasternal to the anterior axillary line and will be divided into upper and lower halves, from the clavicle to the third intercostal space and from the third to the diaphragm. The lateral area (zone 2) will be delineated from the anterior to the posterior axillary line and was divided into upper and basal halves. The posterior area (zone 3) will be considered as the zone beyond the posterior axillary line. The sum of B-lines on each scanning site (0: absence; 1: B7 lines: multiple B-lines 7 mm apart; 2: B3 lines: multiple B 3 mm apart; 3: consolidation) yields a score from 0 to 36(10) score for the ventilated lung is only from 0-18.

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Hosny, MD, Principal Investigator — Kasr Al-Ainy Faculty of Medicine
Locations (1):
- Kasr Al-Ainy faculty of medicine. Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No